CLINICAL TRIAL: NCT05840783
Title: Comparative Evaluation of Postoperative Pain After Using Endoactivator, Side Vented and Open Ended Endodontic Needles as Final Irrigation Protocols During Root Canal Treatment
Brief Title: Evaluation of Post Operative Pain After Sonic Activation and Different Irrigation Needles During Root Canal Treatment
Acronym: Endoactivator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Armed Forces Institute of Dentistry, Pakistan (Other)
Responsible Party: Principal Investigator, Ahmed Abdullah, Registrar Operative Dentistry and Endodontics, Armed Forces Institute of Dentistry, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Sonic activation
Record Dates: First submitted 2023-04-05; First posted 2023-05-03 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Post Operative Pain
Keywords: sonic activation; post operative pain; endoactivator; side vented needle; root canal therapy; irrigation
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients to be divided randomly into three groups after fulfilling the Inclusion Criteria, and not told about the specific intervention being done. Care provider/investigator knows which device they are using, while outcomes accessor is also masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Group A - Open-ended needle (Experimental): Open ended needle group. Irrigation in this group shall be done using a conventional open-ended needle during root canal therapy
  Interventions: Device: Open ended needle irrigation
- Group B- side-vented needle (Experimental): Side vented needle group. Irrigation in this group shall be done using a 30G side-vented needle during root canal therapy
  Interventions: Device: side vented needle irrigation
- Group C- Endoactivator (Experimental): Sonic activation group. In this group, final irrigation during endodontic therapy shall be done using a sonic activation device (Endoactivator)
  Interventions: Device: Sonic activation

INTERVENTIONS:
Device: Open ended needle irrigation — irrigation during root canal shaping and cleaning using an open-ended needle
  Arms: Group A - Open-ended needle
Device: side vented needle irrigation — irrigation during root canal shaping and cleaning using a 30-guage side-vented needle
  Arms: Group B- side-vented needle
Device: Sonic activation — Agitation of root canal irrigation solution with a sonic activation device (Endoactivator).
  Arms: Group C- Endoactivator

SUMMARY:
The study compares the post operative pain after root canal therapy, after using different irrigation protocols. The subjects are divided into 3 groups and different irrigation protocol is used in each group. One group undergoes final irrigation after root canal therapy with a sonic activation device, and in the other two groups, side-vented and open-ended needles are used. Post operative pain is then compared at 8, 24, and 48 hour intervals.

DETAILED DESCRIPTION:
Root canal therapy is a procedure in which inflamed pulp tissue and microorganisms are removed from root canals and pulp chamber, in order to eradicate infection and symptoms. Irrigation is a crucial step of an endodontic therapy and different methods and protocols are used to enhance the efficacy of irrigation. Sonic activation of root canal irrigation agent is one of the effective methods that enhance the outcomes and success rate of endo therapies. It removes the smear layer, bacterial biofilms and debris by acoustic streaming and agitating the irrigant inside root canals. Similarly, irrigation needles also play an important role in endodontic therapy, particularly by improving the delivery of irrigation agent to the apex of a root canal. conventionally, open ended needles have been used for irrigant delivery inside root canal but is not deemed very efficacious as they cannot penetrate deep into canals and cause extrusion of debris beyond the apex. This problem is solved by using side vented needles of smaller gauge (30 G) that leads to better irrigation and prevent extrusion of chemicals and debris outside the root apex.

In this study, the efficacy of all three different irrigation protocols will be compared and assessed based on post-operative pain, measured by Visual Analog Scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unremarkable/ noncontributory medical history
2. Healthy persons between the ages of 18 and 60 years
3. Maxillary and mandibular molar teeth diagnosed with symptomatic irreversible pulpitis.
4. Patients not having taken any medication for 12 hours before treatment
5. No allergies to the drugs or dental material being used in the treatment

Exclusion Criteria:

1. Patients who had taken analgesics on anti-inflammatory drugs within the last 12 hours
2. Pregnant women and patients with immunocompromised health state
3. Patients having severe malocclusion associated with traumatic occlusion
4. Teeth with calcified canals
5. Teeth with periapical radiolucency
6. Teeth with root resorption
7. Teeth previously undergone root canal treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-02-04 (Actual); Study Completion 2024-02-04 (Actual)

PRIMARY OUTCOMES:
Post Operative pain assessed by VAS after endodontic therapy | 1 week
  comparative evaluation of post operative pain after using different irrigation devices, using VAS (Visual Analog Scale). It is drawn as a straight line of 10 inches and marked in numbers which show intensity of pain, from 0-10, with 0 being no pain at all to10 being the worst pain imaginable. In detail, it is a scale which shows pain intensity in ascending order and can also be used to analyze the intensity of pain experienced by the patient.
  0: No pain at all 1-3: mild pain 4-6: moderate pain 7-9: severe pain 10: worst pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Athar Ali, BDS, Study Director — Classified Specialist
Locations (1):
- Armed Forces Institute of dentistry, Rawalpindi, Punjab Province, Pakistan

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-02-02): https://cdn.clinicaltrials.gov/large-docs/83/NCT05840783/Prot_SAP_ICF_000.pdf